CLINICAL TRIAL: NCT00412542
Title: A Phase II Trial of Combination Therapy With Thalidomide and CPT-11 in Patients With Recurrent Anaplastic Gliomas or Glioblastoma Multiforme
Brief Title: Thalidomide and Temozolomide or Camptothecin-11 (CPT-11) in Patients With Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM02-595
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Glioblastoma Multiforme; Glioma
Keywords: Glioblastoma Multiforme; Glioma; Thalidomide; Thalomid; CPT-11; Irinotecan; malignant glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Thalidomide; Irinotecan; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide + CPT-11 (Experimental): Oral Thalidomide 100 mg daily for 8 weeks + CPT-11 125 mg/m^2 by vein weekly over 90 minutes for 4 weeks, followed by 2 weeks rest.
  Interventions: Drug: Thalidomide; Drug: CPT-11; Procedure: MRI Scan; Procedure: Quantitative Sensory Tests (QST)

INTERVENTIONS:
Drug: Thalidomide — 100 mg PO (by mouth) daily for 8 weeks
  Other Names: Thalomid
Drug: CPT-11 — 125 mg/m^2 by vein weekly over 90 minutes for 4 weeks, followed by 2 weeks rest
  Other Names: Irinotecan
Procedure: MRI Scan — Dynamic MRI scan with dye injection through vein, every 6 weeks
  Other Names: Magnetic Resonance Imaging; MR
Procedure: Quantitative Sensory Tests (QST) — QST, every 12 weeks, to check for any nerve problems that may be present before starting treatment; by touching a small machine tests are done on feeling of touch, vibration, and temperature.

SUMMARY:
Objectives:

1.1 To determine the efficacy, as measured by 6 month progression-free survival, of therapy with thalidomide combined with CPT-11 in the treatment of patients with recurrent and/or progressive malignant gliomas.

1.2 To determine the rate of measureable clinical response in patients treated with Thalidomide and CPT-11.

1.3 To determine Thrombotic thrombocytopenic purpura (TTP), overall survival and unexpected toxicity of Thalidomide and CPT-11 used in recurrent malignant gliomas.

1.4 To determine changes in dynamic magnetic resonance imaging (MRI) as a surrogate marker for treatment effect.

DETAILED DESCRIPTION:
Thalidomide is a drug that interferes with the growth of blood vessels. Thalidomide may help to decrease the blood supply in the tumor and make it unable to grow. CPT-11 is a drug that was designed to stop cancer cells from dividing.

All participants will take thalidomide capsules by mouth every evening at bedtime. You will begin with 1 capsule every night for the first week then increase to 2 capsules every night for a week and then 3 capsules a night for the third week. After that, you will increase the dose to 4 capsules each night for the rest of the study. The dosages may be adjusted if you experience any severe side effects.

In addition to thalidomide, you will receive treatment with CPT-11 through a continuous injection into a vein over 90 minutes once a week for 4 weeks followed by 2 weeks of rest from the drug. This 6 week period is called a course of therapy. The courses of therapy will be repeated as long as the disease is responding to treatment for up to 2 years.

THIS IS AN INVESTIGATIONAL STUDY. Both drugs are commercially available. Thalidomide and CPT-11 are FDA approved for the treatment of some cancers. The combination of these drugs is investigational.

Up to 78 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Is there an age limit? No

Inclusion Criteria:

1. Patients with histologically proven supratentorial malignant primary gliomas (Glioblastoma multiforme (GBM), Gliosarcoma (GS) Anaplastic astrocytoma (AA), Anaplastic oligodendroglioma (AO), mixed anaplastic glioma (MAG)) will be eligible for this protocol.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan after radiation therapy.
3. Patients in the GBM stratum may have had treatment for no more than 2 prior relapses; for the AA stratum, there is no limitation for the number of relapses provided all other eligibility criteria particularly the functional status are met.
4. All patients must sign an informed consent.
5. The baseline on-study MRI should be performed within 14 days prior to registration and on a stable or decreasing steroid dosage.
6. Patients having undergone recent resection of recurrent or progressive tumor will be eligible.
7. Patients must have a life expectancy > 8 weeks.
8. Patients must have a Karnofsky performance status of >= 70
9. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count). Patients who receive either Temozolomide or CPT-11 for non-therapeutic purposes (such as presurgically for obtaining pharmacology data for the agent) will be eligible for study entry provided they have recovered from the toxic effects of the agent if any.
10. Patients must have adequate bone marrow function (Absolute neutrophil count (ANC)> 1,500/mm3 and platelet count of > 100,000/mm3), adequate liver function (alanine aminotransferase (ALT or SGPT) and alkaline phosphatase <2 times normal, bilirubin <1.5 mg/dl), and adequate renal function (blood urea nitrogen (BUN) and creatinine <1.5 times institutional normal) prior to starting therapy.
11. Patients must not be pregnant and must practice adequate contraception during the study and for 2 months after participation in study.

Exclusion Criteria:

1. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
2. Patients must not have: a) active infection b) disease that will obscure toxicity or dangerously alter drug metabolism c) serious intercurrent medical illness. d) prior recurrence with CPT-11 (for the CPT-11 + Thalidomide arm) (prior treatment with thalidomide is permitted). e) grade 2 or higher peripheral neuropathy. Patients who have received Temozolomide or CPT-11 for non-therapeutic purposes (for eg., as part of a pharmacology study without therapeutic intent) will remain eligible for enrollment into the study.
3. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MDACC over the past year is as follows: American Indian or Alaskan Native - 0 Asian or Pacific Islander - <2% Black, not of Hispanic Origin - 3% Hispanic - 6% White, not of Hispanic Origin - 88% Other or Unknown - 2% Total-100%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay K. Puduvalli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 13, 2003 to October 22, 2008. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 78 participants enrolled, three (3) were considered not evaluable.
Groups:
- Glioblastoma Multiforme: Thalidomide + CPT-11; Anaplastic Gliomas: Thalidomide + CPT-11: Oral Thalidomide 100 mg daily for 8 weeks + CPT-11 125 mg/m^2 by vein weekly over 90 minutes for 4 weeks, followed by 2 weeks rest.
Period: Overall Study
Arm/Group | Glioblastoma Multiforme: Thalidomide + CPT-11 | Anaplastic Gliomas: Thalidomide + CPT-11
Started | 33 | 45
Completed | 33 | 42
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Not Eligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioblastoma Multiforme: Thalidomide + CPT-11 | Anaplastic Gliomas: Thalidomide + CPT-11 | Total
Number analyzed (Participants) | 33 | 45 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 41 | 72
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 19 | 27
  Male | 25 | 26 | 51
Region of Enrollment [Number; unit: participants]
  United States | 33 | 45 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Progression Free at 6 Months With Malignant Gliomas
Description: Progression-free Survival (PFS) measured as number of participants that are alive and progression-free at 6 months.
Time Frame: 6 Months
Population: 7 participants enrolled were not evaluated as they were evaluable for toxicity only (not having completed the first cycle/clinical decline/etc.).
Measure: Number; unit: participants
Groups:
- Participants With Recurrent Malignant Gliomas: The endpoints combined results of all strata (Arm 1 of Glioblastoma Multiforme: Thalidomide + CPT-11 and Arm 2 of Anaplastic Gliomas: Thalidomide + CPT-11).
Arm/Group | Participants With Recurrent Malignant Gliomas
Number analyzed (Participants) | 68
participants | 24

ADVERSE EVENTS:
Time Frame: 4 years and 11 months
Groups:
- Patients With Recurrent Malignant Gliomas: The endpoints combined results of all strata
Arm/Group | Patients With Recurrent Malignant Gliomas
Serious Adverse Events (participants affected / at risk) | 35/75
Other Adverse Events (participants affected / at risk) | 65/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Recurrent Malignant Gliomas (N=75)
Thrombus pulmonary embolus (Vascular disorders) | 5 (5)
Seizure (Nervous system disorders) | 8 (11) — Patient was admitted overnight for Grade 3 seizure, unlikely related
Nausea (Gastrointestinal disorders) | 3 (3) — Patient was admitted for Grade 2 nausea, possibly related
Vomiting (Gastrointestinal disorders) | 3 (4) — Patient admitted for Grade 2 vomiting, possibly related
Diarrhea (Gastrointestinal disorders) | 9 (10) — Patient admitted for Grade 2 diarrhea, possibly related
Ataxia (Nervous system disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Cerebral edema (Nervous system disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) — Of the 6 deaths reported, 3 were directly related to disease progression of malignant gliomas. The other 3 were due to complications of other events
Dehydration (Gastrointestinal disorders) | 5 (6)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Thrombus - deep vein thrombosis (Vascular disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Elevated ALT (Investigations) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Musculo-skeletal leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Pneumonia (Infections and infestations) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3)
Subdural fluid collection (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Recurrent Malignant Gliomas (N=75)
Abdominal cramping (Gastrointestinal disorders) | 9 (18)
Acne (Skin and subcutaneous tissue disorders) | 12 (17)
Alkaline Phosphatase increased (Investigations) | 11 (18)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13)
ALT increased (Investigations) | 17 (40)
Anemia (Blood and lymphatic system disorders) | 5 (11)
Anorexia (Gastrointestinal disorders) | 22 (25)
AST elevated (Investigations) | 12 (19)
Ataxia (Nervous system disorders) | 6 (9)
Bicarbonate sodium, low (Investigations) | 16 (30)
Bilirubin elevated (Investigations) | 5 (5)
Blurred vision (Eye disorders) | 12 (19)
Bruising (without thrombocytopenia) (Skin and subcutaneous tissue disorders) | 5 (5)
BUN elevated (Investigations) | 12 (20)
Cholesterol elevated (Investigations) | 11 (11)
Cognitive disturbance (Nervous system disorders) | 8 (8)
Confusion (Psychiatric disorders) | 16 (22)
Constipation (Gastrointestinal disorders) | 46 (91)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (33)
CPK elevated (Investigations) | 4 (5)
Creatinine elevated (Investigations) | 9 (11)
Cushingoid (Endocrine disorders) | 11 (11)
Dehydration (Gastrointestinal disorders) | 14 (16)
Diarrhea (Gastrointestinal disorders) | 46 (171)
Dizziness (Nervous system disorders) | 32 (55)
Dry mouth (General disorders) | 9 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (17)
Dysphasia (Nervous system disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (21)
Edema (General disorders) | 31 (42)
Elevated chloride (Investigations) | 18 (38)
Elevated CO2 (Investigations) | 14 (27)
Elevated AST (Investigations) | 6 (8)
Fatigue (General disorders) | 63 (143)
Fever without neutropenia (General disorders) | 11 (16)
Gait/walking (Nervous system disorders) | 31 (37)
Anemia/decreased hemoglobin (Blood and lymphatic system disorders) | 57 (195)
Hyperglycemia (Metabolism and nutrition disorders) | 49 (130)
Hyperuricemia (Investigations) | 7 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 (53)
Hypocalcemia (Metabolism and nutrition disorders) | 21 (57)
Hypokalemia (Investigations) | 24 (47)
Hypomagnesium (Investigations) | 13 (16)
Hyponatremia (Investigations) | 19 (34)
Hypophosphatemia (Investigations) | 24 (56)
Hypotension (Vascular disorders) | 9 (10)
Incontinence, urinary (Renal and urinary disorders) | 8 (8)
Infection (Infections and infestations) | 23 (26)
Insomnia (General disorders) | 18 (24)
Leukopenia (Blood and lymphatic system disorders) | 65 (315)
Low protein (Investigations) | 15 (21)
Lymphopenia (Blood and lymphatic system disorders) | 52 (284)
Memory Impairment (Nervous system disorders) | 26 (29)
Mood alteration (Psychiatric disorders) | 18 (20)
Mucositis (Gastrointestinal disorders) | 10 (13)
Muscle weakness lower extremity (Musculoskeletal and connective tissue disorders) | 25 (36)
Muscle weakness facial (Musculoskeletal and connective tissue disorders) | 6 (7)
Muscle weakness left or right sides (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle weakness generalized (Musculoskeletal and connective tissue disorders) | 15 (21)
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 38 (119)
Neuropathy motor (Nervous system disorders) | 11 (14)
Neuropathy sensory (Nervous system disorders) | 35 (52)
Neutrophils, absolute count (Blood and lymphatic system disorders) | 55 (249)
Pain, abdominal (Gastrointestinal disorders) | 17 (34)
Pain, back (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain, chest (non cardiac) (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain, extremity (Musculoskeletal and connective tissue disorders) | 9 (18)
Pain, headache (Nervous system disorders) | 39 (75)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (52)
Pyramidal tract dysfunction (Nervous system disorders) | 19 (27)
Seizure (Nervous system disorders) | 25 (48)
Somnolence (Nervous system disorders) | 20 (25)
Speech impairment (Nervous system disorders) | 19 (28)
Tremors (Nervous system disorders) | 18 (22)
Urinary frequency (Renal and urinary disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 22 (57)
Weight gain (Metabolism and nutrition disorders) | 10 (12)
Weight loss (Metabolism and nutrition disorders) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes